CLINICAL TRIAL: NCT06152848
Title: The SAM Project: Science Against Malnutrition Project
Status: Recruiting | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Medical Doctor, PhD, Professor, Federico II University
Other Study IDs: 2/2023
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients affected by malnutrition: Patients affected by malnutrition due to deficiency or excess
  Interventions: Other: Data and samples collection
- Sex- and age- matched healthy controls: Sex- and age- matched healthy controls not affected by any pathology and/or malnutrition due to deficiency or excess
  Interventions: Other: Data and samples collection

INTERVENTIONS:
Other: Data and samples collection — Collection of clinical, anamnestic and lifestyle data; collection of faecal, blood and saliva samples

SUMMARY:
The latest data from the World Health Organization (WHO) shows that malnutrition in all its forms affects over 2.5 billion people globally. This condition is constantly increasing and affects the entire population, from childhood to the elderly. Malnutrition in all its forms negatively impacts the quality of life of patients affected and increases the risk of morbidity and mortality, as well as healthcare costs. Considering the complexity and multifactorial nature of malnutrition, the integration of multi-omics data obtained from analyzes with high-throughput technologies such as epigenomics, metagenomics, metabolomics, could benefit the prediction and evaluation of prognosis and/or response to specific treatments; this could pave the way for personalized precision medicine interventions for patients suffering from malnutrition. The SAM study aims to characterize malnutrition through the identification of specific biomarkers of the condition with the aim of developing innovative prevention and treatment programs.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian ethnicity;
* both sexes;
* age between 0 and 85 years;
* affected by malnutrition due to deficiency or excess in association with other patology and sex- and age-matched healthy controls not affected by malnutrition due to deficiency or excess and any pathology
* Written informed consent

Exclusion Criteria:

* Non-Caucasian ethnicity;
* Age > 85 years.

Ages: 0 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1000 patients affected by malnutrition due to deficiency or excess, associated with at least one of the pathological conditions(small for gestational age; metabolic syndrome; type 1 diabetes mellitus; neurological diseases; psychiatric; chronic infectious diseases; oncological pathologies; gastrointestinal diseases; cardiovascular diseases; kidney disease; lung pathologies) aged 0-85 years (50% male) and 1000 sex- and age- matched healthy controls not affected by any pathology and/or malnutrition due to deficiency or excess.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2026-07-24 (Estimated); Study Completion 2026-07-24 (Estimated)

PRIMARY OUTCOMES:
Characterization of malnutrition through the identification of specific biomarkers of the condition. | 36 months
  Data and samples analyses
Untargeted microRNA expression profile in blood samples | 36 months
  TruSeq Small RNA Sample Preparation Kit (Illumina)
Plasmatic extracellular vesicles | 36 months
  A transmission electron microscope will be used to analyze the morphology of extracellular vesicles and the total protein concentration of the extracellular vesicles will be measured with a Bradford assay and the quantitation of specific membrane proteins and specific intracellular proteins (Heat-Shock Proteins/HSP) will be carried out by ELISA.
Metagenomic analysis of fecal samples | 36 months
  Shotgun analysis
Metabolomicanalysis of fecal samples | 36 months
  Gas chromatography-mass spectrometry
Untargeted microRNA expression profile in saliva samples | 36 months
  TruSeq Small RNA Sample Preparation Kit (Illumina)
Salivary extracellular vesicles | 36 months
  A transmission electron microscope will be used to analyze the morphology of extracellular vesicles and the total protein concentration of the extracellular vesicles will be measured with a Bradford assay and the quantitation of specific membrane proteins and specific intracellular proteins (Heat-Shock Proteins/HSP) will be carried out by ELISA.
Metagenomic analysis of salivary samples | 36 months
  Shotgun analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Traslational Medical Science - University of Naples Federico II, Naples, Italy